CLINICAL TRIAL: NCT00827463
Title: The Early Detection of Anaemia During the Maternity Decreases the Anaemia at the End of the Maternity.
Brief Title: Early Detection of Anaemia During the Maternity
Acronym: anémie
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: I08009
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2009-09

CONDITIONS: Anemia
Keywords: aneamia; aneamia during the maternity
MeSH Terms: conditions — Anemia | interventions — Iron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NFS and iron in the first quater (Experimental): first arm: dosage NFS and iron during the beginning of the pregnancy then in the sixth month of pregnancy then in th delivery.
  Interventions: Biological: dosage of the NFS and iron
- No NFS and iron in the first quater (Experimental): second arm: dosage NFS and iron during the sixth month of pregnancy then in th delivery. No dosage of NFS and iron during the beginning of the pregnancy
  Interventions: Biological: dosage of the NFS and iron

INTERVENTIONS:
Biological: dosage of the NFS and iron — a blood test will be made.

SUMMARY:
Estimate the efficiency of a strategy of premature screening of the maternal anaemia during the first quarter of pregnancy versus the usual strategy of screening of the anaemia during the sixth month.

DETAILED DESCRIPTION:
A part of the patient will have a NFS and dosage of the cast-iron, during the results of the beginning of the pregnancy at the first quarter.

The other part of the patients will have a NFS and at the first quater of the pregnancy.

All the patient will have a NFS at the results of the sixth month of the pregnancy.

A NFS will be done during the results at the end of the pregnancy like we do now.

Then a NFS at 48 hours after the birth. A treatment with iron will be done and according to the results

ELIGIBILITY:
Inclusion Criteria:

* Every patient followed at the HME at the beginnig of the pregnancy

Exclusion Criteria:

* pregnency women who don't speak french
* pregnancy women affected by béta thalassemia
* pregnancy woman having had a périconceptionnel treatment against the anaemia

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
primary outcomes: is the rate of heamophilia at the end of the pregnancy. | six months

SECONDARY OUTCOMES:
Secondary outcomes: - the percent of treatment of intravenous irons during the pregnancy and the following layers. - the percent of transfusion and the following layers. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Vincelot anne, MD, Principal Investigator — Limoges UH
Locations (1):
- CHU limoges, Limoges, Limousin, France